CLINICAL TRIAL: NCT03143270
Title: A Multicenter Pilot Study of Nivolumab With Drug Eluting Bead Transarterial Chemoembolization in Patients With Advanced Hepatocellular Carcinoma
Brief Title: A Study to Test the Safety and Feasibility of Nivolumab With Drug Eluting Bead Transarterial Chemoembolization in Patients With Liver Cancer
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-087
Record Dates: First submitted 2017-05-01; First posted 2017-05-08 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Liver Cancer
Keywords: nivolumab; deb-TACE; 17-087
MeSH Terms: conditions — Liver Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1, deb-TACE + Nivolumab (Experimental): 3 eligible participants will undergo deb-TACE on Day 0 (+/- 5 days). Two weeks after deb-TACE, participants will begin nivolumab every two weeks for up to one year. If no participants experience a dose limiting toxicity (DLT), or 1 of 6 participants experiences a DLT, a new group of participants will be enrolled into Cohort 2.
  Interventions: Drug: Drug Eluting Bead Transarterial Chemoembolization; Drug: Nivolumab
- Cohort 2, deb-TACE + Nivolumab (Experimental): 3 eligible participants will undergo deb-TACE on Day 0 (+/- 5 days). Participants will receive nivolumab every two weeks for up to one year, starting 4 weeks prior to deb-TACE (week -4). Participants in this cohort will not receive nivolumab on the day of deb-TACE. If no participants experience a DLT in the initial group of 3 participants or if 1 of 6 participants experiences a DLT, a new group of participants will be enrolled into Cohort 3.
  Interventions: Drug: Drug Eluting Bead Transarterial Chemoembolization; Drug: Nivolumab
- Cohort 3, deb-TACE + Nivolumab (Experimental): 3 eligible participants will undergo deb-TACE on Day 0 (+/- 5 days). Nivolumab will be dosed every two weeks starting 4 weeks prior to deb-TACE (Week 4) and continue every 2 weeks for up to one year. If no participants experience a DLT in the initial group of 3 participants, an additional 3 participants will be added to confirm safety. If less than or equal to 1 of 6 participants experiences a DLT, this will be considered the optimal schedule.
  Interventions: Drug: Drug Eluting Bead Transarterial Chemoembolization; Drug: Nivolumab

INTERVENTIONS:
Drug: Drug Eluting Bead Transarterial Chemoembolization — Hepatic embolization will occur on Day 0 of the study for all cohorts. On the day of the procedure, baseline angiography including celiac and superior mesenteric angiography will be performed to delineate arterial anatomy and blood supply to the tumor. After the entire dose has been used, the embolized vessels will be re-catheterized and embolized to stasis with Bead Block beginning with 100-300 micron spheres and using a maximum of 10 cc of any given size per vessel before moving to the next size microsphere.
  Other Names: deb-TACE
Drug: Nivolumab — All participants will receive at a flat dose of 240 mg IV q 12 weeks for up to one year. In cohort 1, participants will begin nivolumab two weeks (+/- 5 days) after deb-TACE every two weeks. In cohort 2, participants will begin nivolumab every 2 weeks for 1 year and undergo deb-TACE 4 weeks after the initiation of nivolumab (+/- 5 day). Nivolumab will not be dosed on the day of embolization in this cohort. In cohort 3, nivolumab will be dosed every two weeks starting 4 weeks (+/- 5 days) prior to deb-TACE and continue every 2 weeks for up to one year. Nivolumab will be dosed on the day of embolization in this cohort. It will be administered before the deb-TACE procedure.

SUMMARY:
The purpose of the study is to find out the effects of using nivolumab with Drug Eluting Bead Transarterial Chemoembolization (deb-TACE) in the treatment of liver cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over at the time of consent
* Histology and/or cytology confirmed HCC per the enrolling institution. Subjects in Cohort 1 are permitted to enroll w ithout confirmation of HCC as long as imaging LiRADs criteria are met and a biopsy is scheduled prior to or the day of the deb-TACE procedure. HCC confirmation must be completed prior to initiation of nivolumab for all cohorts. If a patient is found to not have confirmed HCC, they w ill be removed from the study.
* Measurable disease per RECIST v1.1
* Disease not amenable to curative or transplant surgery (BCLC Stage B); disease must be reviewed by members of disease management team at the local enrolling institution and be amenable to deb-TACE. For the dose escalation and the expansion, regional lymphadenopathy and sub-centimeter pulmonary nodules are allowed as well as segmental portal vein involvement.
* ECOG Performance status 0 or 1
* Child-Pugh Class A
* Child-Pugh Scoring Note: PI INR <1.7 is not required for patients on anticoagulation agents. Patients who are being therapeutically anticoagulated with an agent such as Coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists
* Adequate bone marrow, hepatic, and renal function defined as:

  * Platelet count ≥ 75,000/mm3
  * Absolute neutrophil count ≥ 1,000/mm3
  * Hemoglobin ≥ 9 g/dL
  * Total bilirubin < 3.0 × ULN (upper limit of normal)
  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 5 × ULN
  * Albumin ≥ 2.8 g/dL
  * Serum creatinine ≤ 1.5 mg/dL or calculated creatinine clearance ≥ 40 mL/min as determined by the Cockcroft-Gault equation
* Suppression of HBV (≤ 100 IU/mL by HBV PCR) with antivirals per the local standard of care if prior or current HBV exposure or infection.
* Active HCV infection without treatment is permitted. Concomitant treatment of HCV is not permitted on this study.

Exclusion Criteria:

* Vascular invasion or extrahepatic spread
* History of liver allograft; prior hepatic resection is allowed.
* Prior embolization and/or ablation is allowed as long as the patient has progressed with a new RECIST measurable lesion
* Contraindication to angiography/embolization procedure based on judgment of the treating investigator.
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* A history of a severe contrast allergy (.i.e. anaphylaxis) not controlled with premedication
* Patients should be excluded if they have a condition requiring chronic systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Patients with contrast allergies who can tolerate contrast with corticosteroid premedication are not excluded.
* An active, known or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
* Subjects with history of another primary cancer, with the exception of: a) curatively resected non-melanoma skin cancer; b) curatively treated cervical carcinoma in situ; or c) other primary solid tumor with no known active disease present that in the opinion of the investigator will not affect patient outcome in the setting of current HCC diagnosis.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results
* Women of childbearing potential (WOCBP) or sexually active men must use appropriate method(s) of contraception.

  * Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception while on study treatment. WOCBP should use an adequate method to avoid pregnancy during study treatment and for 5 months (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug
  * Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception during study treatment and for a period of 7 months after the last dose of investigational product
  * Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile, as well as azoospermic men do not require contraception
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of nivolumab. Elevated HCG for other explained and documented reasons is allowed.
* Lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 12 months
  The percentage of subjects who experience toxicity at each schedule will be calculated. Frequencies of toxicities will be tabulated according to the NCI CTCAE scale (version 4.03).

CONTACTS AND LOCATIONS:
Overall Officials: James Harding, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Abramson Cancer Center at University of Pennsylvania Medical Center, Philadelphia, Pennsylvania

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/